CLINICAL TRIAL: NCT05054959
Title: Induction Versus Consolidation Chemotherapy in Total Neoadjuvant Therapy of Localy Advanced Rectal Cancer With High Risk of Recurrence (ICONA Study)
Brief Title: Consolidation Versus Induction Chemotherapy in Total Neoadjuvant Therapy of Rectal Cancer With High Risk for Recurrence
Acronym: ICONA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Principal Investigator, Violeta Kaluza, Institute of Oncology Ljubljana, Institute of Oncology Ljubljana
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KME 0120-214/2021/3
Record Dates: First submitted 2021-09-19; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Locally Advanced Rectal Cancer
Keywords: rectal cancer; total neoadjuvant therapy; induction chemotherapy; consolidation chemotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Consolidation Chemotherapy; Induction Chemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- consolidation chemotherapy (Experimental): chemoradiation: intensity-modulated irradiation technique with simultaneous integrated boost to the tumor (IMRT-SIB) or with volumetric modulated arc therapy (VMAT) with simultaneous integrated boost (VMAT-SIB) to the total tumor dose of 46.2 Gy in T1-3 tumors and 48.4 Gy in T4 tumors in 22 fractions with concomitant CT with capecitabine (dosage: 825 mg / m2 / 12 h per os continuously from the first to the last day of irradiation).
  6 cycles of CAPOX chemotherapy. One cycle of CAPOX CT lasts 3 weeks and consists of capecitabine 1000 mg / m2 / 12h per os for 1-14 days and oxaliplatin 130 mg / m2 intravenously in a two-hour infusion on day 1.
  Interventions: Other: consolidation chemotherapy
- induction chemotherapy (Active Comparator): 4 cycles of induction CAPOX chemotherapy. One cycle of CAPOX CT lasts 3 weeks and consists of capecitabine 1000 mg / m2 / 12h per os for 1-14 days and oxaliplatin 130 mg / m2 intravenously in a two-hour infusion on day 1.
  Chemoradiation:intensity-modulated irradiation technique with simultaneous integrated boost to the tumor (IMRT-SIB) or with volumetric modulated arc therapy (VMAT) with simultaneous integrated boost (VMAT-SIB) to the total tumor dose of 46.2 Gy in T1-3 tumors and 48.4 Gy in T4 tumors in 22 fractions with concomitant CT with capecitabine (dosage: 825 mg / m2 / 12 h per os continuously from the first to the last day of irradiation).
  2 cycles of consolidation CAPOX chemotherapy.
  Interventions: Other: induction chemotherapy

INTERVENTIONS:
Other: consolidation chemotherapy — 6 cycles CAPOX after chemoradiotherapy
  Arms: consolidation chemotherapy
Other: induction chemotherapy — 4 cycles CAPOX before and 2 cycles CAPOX after chemoradiotherapy
  Arms: induction chemotherapy

SUMMARY:
The purpose of the study is to identify the most promising sequence of modalities in total neoadjuvant treatment of localy advanced rectal cancer with high risk of recurrence

DETAILED DESCRIPTION:
International recommendations for the treatment of LARC with a high risk of disease recurrence are inconsistent, regarding TNT. In Germain randomised study more pCR were achieved with consolidation chemotherapy. We will compare our standard approach (induction plus consolidation CT) with consolidation CT.

ELIGIBILITY:
Inclusion Criteria:- histologically proven rectal adenocarcinoma

* no distant metastases on CT scan (M0 disease)
* at least one high risk factor for disease recurrence identified on MR imaging:

  * T4 tumor (cT4)
  * N2 disease (cN2)
  * extramural venous invasion (cEMVI+)
  * positive lateral lymph nodes
  * distance of tumor to mesorectal fascia or positive lymph nodes is 1 mm or less (cMRF+)
* capacity for informed consent
* willingness to attend regular check-ups during and after treatment

Exclusion Criteria:history of previous irradiation in the pelvic area

* absolute contraindications for MR imaging
* distant metastases cannot be reliably excluded
* synchronous cancer
* chronic inflammatory bowel disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
complete remission rate | 2 weeks after completiton of TNT
  The proportion of complete responses will be defined as the sum of the proportions of pCR in operated patients and cCR in non-operated patients.

SECONDARY OUTCOMES:
Overall survival | after 3 years of follow-up
  time from randomization to death
Survival without recurrence of the disease | after 3 years of follow-up
  time from the end of treatment (in the case of cCR) or from radical surgery to death or recurrence of the disease - whichever comes first.
Disease free survival | after 3 years of follow-up
  the time from the end of treatment (in the case of cCR) or surgery to the recurrence of disease, the onset of new cancer, death from cancer or other causes
local control | after 3 years of follow-up
  the time from the end of the treatment (in the case of cCR) or surgery to local recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Vaneja Velenik, PD, Principal Investigator — Institute of Oncology Ljubljana
Locations (1):
- Institute of Oncology, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cercek A, Goodman KA, Hajj C, Weisberger E, Segal NH, Reidy-Lagunes DL, Stadler ZK, Wu AJ, Weiser MR, Paty PB, Guillem JG, Nash GM, Temple LK, Garcia-Aguilar J, Saltz LB. Neoadjuvant chemotherapy first, followed by chemoradiation and then surgery, in the management of locally advanced rectal cancer. J Natl Compr Canc Netw. 2014 Apr;12(4):513-9. doi: 10.6004/jnccn.2014.0056. PMID 24717570
- [Background] Tuta M, Boc N, Brecelj E, Peternel M, Velenik V. Total neoadjuvant therapy vs standard therapy of locally advanced rectal cancer with high-risk factors for failure. World J Gastrointest Oncol. 2021 Feb 15;13(2):119-130. doi: 10.4251/wjgo.v13.i2.119. PMID 33643528
- [Background] Tuta M, Boc N, Brecelj E, Omejc M, Anderluh F, Ermenc AS, Peressutti AJ, Oblak I, Krebs B, Velenik V. Total neoadjuvant treatment of locally advanced rectal cancer with high risk factors in Slovenia. Radiol Oncol. 2019 Oct 25;53(4):465-472. doi: 10.2478/raon-2019-0046. PMID 31652124
- [Background] Fokas E, Allgauer M, Polat B, Klautke G, Grabenbauer GG, Fietkau R, Kuhnt T, Staib L, Brunner T, Grosu AL, Schmiegel W, Jacobasch L, Weitz J, Folprecht G, Schlenska-Lange A, Flentje M, Germer CT, Grutzmann R, Schwarzbach M, Paolucci V, Bechstein WO, Friede T, Ghadimi M, Hofheinz RD, Rodel C; German Rectal Cancer Study Group. Randomized Phase II Trial of Chemoradiotherapy Plus Induction or Consolidation Chemotherapy as Total Neoadjuvant Therapy for Locally Advanced Rectal Cancer: CAO/ARO/AIO-12. J Clin Oncol. 2019 Dec 1;37(34):3212-3222. doi: 10.1200/JCO.19.00308. Epub 2019 May 31. PMID 31150315
- [Background] Golo D, But-Hadzic J, Anderluh F, Brecelj E, Edhemovic I, Jeromen A, Omejc M, Oblak I, Secerov-Ermenc A, Velenik V. Induction chemotherapy, chemoradiotherapy and consolidation chemotherapy in preoperative treatment of rectal cancer - long-term results of phase II OIGIT-01 Trial. Radiol Oncol. 2018 Sep 11;52(3):267-274. doi: 10.2478/raon-2018-0028. PMID 30210040
- [Background] But-Hadzic J, Anderluh F, Brecelj E, Edhemovic I, Secerov-Ermenc A, Hudej R, Jeromen A, Kozelj M, Krebs B, Oblak I, Omejc M, Vogrin A, Velenik V. Acute Toxicity and Tumor Response in Locally Advanced Rectal Cancer After Preoperative Chemoradiation Therapy With Shortening of the Overall Treatment Time Using Intensity-Modulated Radiation Therapy With Simultaneous Integrated Boost: A Phase 2 Trial. Int J Radiat Oncol Biol Phys. 2016 Dec 1;96(5):1003-1010. doi: 10.1016/j.ijrobp.2016.08.031. Epub 2016 Aug 31. PMID 27727065